CLINICAL TRIAL: NCT06454253
Title: the Ethics Committee of the First Affiliated Hospital of Nanchang University
Brief Title: Short- and Long-term Outcomes of Robotic vs Laparoscopic Right Colon Cancer: a 10-year Single-center Retrospective Study
Status: Completed | Type: Observational
Sponsor: Taiyuan Li (Other)
Responsible Party: Sponsor-Investigator, Taiyuan Li, the First Affiliated Hospital of Nanchang University, Nanchang University
Organization: Nanchang University (Other)
Other Study IDs: IIT2023015
Record Dates: First submitted 2024-05-29; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Robotic; Laparoscopic; Colon Cancer; Long-term Outcomes; Short-term Outcomes
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- robot-assisted right colon group: Robot assisted radical surgery for right colon cancer
  Interventions: Device: Da Vinci Robot Surgical System
- laparoscopic-assisted right colon group: Laparoscopic assisted radical surgery for right colon cancer
  Interventions: Device: Da Vinci Robot Surgical System

INTERVENTIONS:
Device: Da Vinci Robot Surgical System — Performing surgery on right colon cancer patients using the da Vinci robotic surgical system or laparoscopic surgical system
  Other Names: Laparoscopic surgical system

SUMMARY:
The goal of this observational study is to evaluate the short-term outcomes and long-term outcomes of robot-assisted right colon group for cancer compared to laparoscopic-assisted right colon group. This is a large sample study based on ten years of clinical data. The main question it aims to answer is: What are the advantages of da Vinci robot right hemicolectomy compared to laparoscopic right hemicolectomy, and is there a difference in long-term efficacy between the two methods.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is highly prevalent worldwide. In China, CRC ranks high among the population of men and women with cancer. The incidence and mortality rates of CRC are rising quickly in developing countries, and it is the fourth most deadly cancer in the world. In particular, the right colon cancer (RCC) is continuously growing in China, and the early symptoms of RCC are not typical. one of the most useful ways for RCC is surgical is a surgical operation. Along with the development of minimally invasive surgery, the use of laparoscopy for colon cancer is widely accepted and has become one symbolic surgical technology. Studies have demonstrated that laparoscopic colonic surgery is related to reduced pain after operation, shorter rehabilitation time, shorter length of hospital stay, reduced the time of ileus after surgery, and reduced surgical site infection.

Nevertheless, laparoscopic surgery also has its shortcoming, including a limited range of motion, slow learning and growth, and physiological tremor cannot be eliminated.The emergence of robots has broken the inherent disadvantage of laparoscopy. It has achieved similar or better results in previous studies. Based on these advantages, robotic surgery has received much attention from the surgeons. With the first robotic surgery in the field of colon cancer was reported in 2002, there are some studies proved the safety and feasibility by using robot,However, most studies with small sample sizes and with cases at a relatively early stage.

Therefore, the purpose of this study is to compare the short-term and long-term outcomes between RARC and LARC in the treatment of right colon cancer in our center.

ELIGIBILITY:
Inclusion Criteria:

1. The age is more than 18 years old and less than or equal to 85 years old
2. No distant metastasis (including pelvic cavity, peritoneum, liver, lung, brain, bone, distant lymph node metastasis, etc.) is judged by ultrasound, CT, PET-CT, etc
3. Preoperative colonoscopy showing that the tumor was located in the ileocecal region, ascending colon, hepatic flexure, or transverse colon with pathology showing malignancy
4. signed informed consent. -

Exclusion Criteria:

1. multiple primary colorectal cancer
2. recurrent right colon cancer
3. preoperative neoadjuvant chemotherapy
4. emergency surgery for intestinal obstruction, bleeding or perforation
5. incomplete data and missing follow-up data. -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The consecutive cases of robotic-assisted or laparoscopic-assisted right colectomy between December 2014 and March 2024. All cases derived from the First Affiliated Hospital of Nanchang University.
Sampling Method: Non-Probability Sample
Enrollment: 1879 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
overall survival | 5 years after surgery
  months
disease-free survival | 5 years after surgery
  months

SECONDARY OUTCOMES:
the rate of postoperative complications | 1 months after surgery
  rate
operative time | Intraoperative
  minutes
estimation of blood loss | Intraoperative
  milliliters
number of retrieved lymph nodes | Intraoperative
  numbers
days after postoperative hospital stay | 1 months after surgery
  days
time to first exhaust | 1 weeks after surgery
  hours
time to liquid diet | 1 weeks after surgery
  hours
the rate of intracorporeal anastomosis | 1 months after surgery
  rate

IPD SHARING:
Plan to Share IPD: Undecided
Access to the database can be obtained from the corresponding author on reasonable request.

DOCUMENTS (1):
  • Study Protocol (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT06454253/Prot_000.pdf